CLINICAL TRIAL: NCT02639273
Title: Effect of Opioid Receptor Modulation on Alcohol Self-Administration and Neural Response to Alcohol Cues in Heavy Drinkers: Role of OPRM1 Gene Variation
Brief Title: Title: Effect of Opioid Receptor Modulation on Alcohol Self-Administration and Neural Response to Alcohol Cues in Heavy Drinkers: Role of OPRM1 Gene Variation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 160037; 16-AA-0037
Record Dates: First submitted 2015-12-23; First posted 2015-12-24 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2025-10-23

CONDITIONS: AUD
Keywords: Alcohol Infusion study; Nalmefene; fMRI; Genetics; NIAAA
MeSH Terms: interventions — nalmefene

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Drug (Experimental): single dose nalmefene
  Interventions: Drug: Nalmefene
- Placebo (Placebo Comparator): single dose placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Nalmefene — Active Drug
  Arms: Drug
Other: Placebo — Single Dose Placebo
  Arms: Placebo

SUMMARY:
Background:

Drugs like nalmefene interfere with opioid receptors. This might reduce drinking. The gene OPRM1 determines opioid receptor functions. Researchers want to see if nalmefene affects people s responses to alcohol cues. They also want to compare how nalmefene affects people with different forms of OPRM1.

Objectives:

To test nalmefene s effects on alcohol self-infusion and responses to alcohol cues. To test the role of different forms of OPRM1 on these effects.

Eligibility:

Healthy heavy drinkers ages 21 60:

Women: over 15 drinks weekly

Men: over 20 drinks weekly

Design:

Participants will be screened with:

Medical history

Physical exam

Heart, blood, and urine tests

Questionnaires

Participants will have three 10-hour visits and one 2-hour follow-up visit. They will take a taxi. Visits are about 1 week apart.

Before visits, participants cannot drink alcohol for 1 day or take medicine for 3 days.

All study visits:

Questionnaires

Heart monitor

Two-hour alcohol session: A needle guides a thin plastic tube into a vein in each arm. One tube receives alcohol. The other draws blood. Participants give themselves alcohol by pressing a button on a computer.

Relaxing at the center until breath alcohol falls below 0.02 percent, or for 3 hours.

Visits 2 and 3:

Swallowing nalmefene or placebo.

One-hour brain MRI: Participants lie on a table with a coil on their head. They press buttons in response to computer cues.

Follow-up visit: participants will discuss their drinking habits.

DETAILED DESCRIPTION:
Previous studies have shown that the opioid receptor modulator nalmefene can reduce heavy drinking among alcoholics. Genetic variation at the micro-opioid receptor gene locus, OPRM1, specifically the A118G polymorphism, is associated with differential subjective responses to alcohol. Further, the A118G polymorphism has been shown to moderate the effect of opioid receptor modulators on alcohol consumption. However, the role of A118G on nalmefene s effectivenes, and the neural substrates underlying nalmefene s therapeutic effect remain to be explored in humans.

Objective: To evaluate the effect of nalmefene on alcohol self-infusion and neural response to alcohol cues in healthy male and female heavy drinkers, and to examine the role of the OPRM1 A118G polymorphism on this effect.

Study population: Participants will be 21-60 year-old male and female heavy drinkers in good health, as determined by medical history, physical exam, and ECG and lab tests. Participants with current Axis-I mood, anxiety or substance use diagnoses, except alcohol dependence, will be excluded. Participants will be divided into 2 genotypic groups: Group 1 (AA) will include participants homozygous for the major 118A allele (118AA genotype), and group 2 (GX) will include participants carrying 1 or 2 copies of the variant 118G allele (118AG or 118GG genotype).

Design: Participants will undergo 3 study sessions. In the first session, participants will complete an intravenous alcohol self-administration (IV-ASA) where they will have an open bar phase to determine their baseline level of alcohol consumption in the laboratory, as well as to obtain data on tolerability and subjective measures of alcohol effects. In the second and third sessions, participants will receive a single dose of either nalmefene or placebo, in counter-balanced order, before completing functional magnetic resonance imaging (fMRI) scans and IV-ASA procedures. The fMRI scans will include a task where participants will see cues that indicate the possibility of earning alcohol rewards to examine the neural substrates involved in processing alcohol cues, and a task designed to measure neural responses during anticipation and processing of aversive events. The difference in alcohol self-infusions between the two sessions will be compared between the two genotypic groups.

Outcome measures: The primary outcome measures are: (1) nalmefene-induced changes in IV alcohol self-administration; (2) nalmefene-induced BOLD signal changes in neural regions associated with alcohol reward processing, including ventral striatum, amygdala, and insula.;Secondary outcome measures include: (1) Nalmefene-induced BOLD signal changes in neural processing of aversive stimuli during fMRI; (2) Genotypic modulation (at the OPRM1 118 location) of nalmefene s effects on primary outcome measures (BOLD signal change during alcohol reward processing and IV alcohol self-administration).

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

Participants will be healthy 21-60 year-old male and female heavy drinkers. An equal number of participants with OPRM 118 AA genotype and those with 1 or 2 copies of the G allele (AG or GG) will be enrolled. Inclusion and exclusion criteria will be evaluated following screening conducted under the NIAAA screening protocol as described below

INCLUSION:

* Male and female participants between 21-60 years of age.
* Male participants must have consumed an average of greater than 14 standard drinks per week, and females must have consumed an average of greater than 7 standard drinks per week during the past 3 months [assessment: 90-day timeline followback (TLFB)completed at screening visit].
* In addition, participants must have on average at least 1 binge drinking day per week during the last 90 days, defined as a day in which 4 or more standard drinks were consumed for females and 5 or more standard drinks were consumed for males. Average number of binge drinking days will be calculated based on total number of binge drinking days from the TLFB (e.g., for 90 days worth of data, participants with a total of 13 or more binge drinking days will be eligible).
* Participants must be willing and able to refrain from using alcohol one day prior to each study, and non-prescription medication for 3 days prior to each visit [assessment: medical history].
* Inclusion criteria for women:

  * Use of adequate method of birth control during the study, if female is sexually active and is not surgically sterilized. Adequate methods of contraception include: use of oral contraceptives; use of barrier method of contraceptive; use of an approved IUD or other long-acting reversible contraceptive (LARC); have a male sexual partner who is surgically sterilized; or have exclusively female sexual partner(s) [assessment: medical history].

EXCLUSION:

* Current or prior history of major medical illness, including CNS, cardiovascular, respiratory, gastrointestinal, hepatic, renal, endocrine, or reproductive disorders [assessment: clinically significant findings on medical history and physical exam, ECG, laboratory tests].
* Participation in any other pharmacological intervention study within 4 months prior to the start of this study [assessment: medical history].
* Positive hepatitis A, B Antigen, or C, or HIV test [assessment: laboratory test].
* An aspartate transaminase (AST) / alanine transaminase (ALT) ratio 3 times greater than the normal limit [assessment: laboratory test].
* Diagnosis of Axis-I anxiety disorders or major depressive disorders in the past 12 months [assessment: SCID interview].
* Lifetime diagnosis of Axis-I bipolar disorders or psychotic disorders [assessment: SCID interview].
* Suicidal ideation in the past 6 months or suicidal behavior in the past 12 months [assessment: Columbia Suicide Severity Rating Scale].
* Current diagnosis of substance use disorder (SUD), other than alcohol use disorder, mild cannabis use disorder (less than 4 criteria), or current SUD in remission. Current smoking or nicotine dependence is not exclusionary [assessment: SCID-IV/SCID-5 interview, FTND].
* Positive result on urine drug screen or breathalyzer test during screening. Positive urine drug screen or breathalyzer reading during more than 1 study visit will result in participant withdrawal from the study [assessment: laboratory tests and breathalyzer test performed at screening or update visit under 14-AA-0181 most proximal to enrollment].
* Currently (i.e., at the time of screening) seeking treatment for alcohol problems or have undergone inpatient or outpatient detoxification or treatment for alcohol problems in the past 6 months. [assessment: medical history and physical exam].
* Lactose intolerance or rare hereditary problems of galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption [assessment: medical history and physical exam].
* Alcohol use:

  * Current or prior history of alcohol-induced flushing reaction, including rapid reddening of the face, rapid heart rate and breathing, and nausea after 1 or 2 drinks [assessment: medical history and physical exam, alcohol flushing questionnaire].
  * History of delirium tremens, hallucinations or seizures related to alcohol withdrawal [assessment: medical history, CIWA-Ar, SCID interview].
* Medication exclusion criteria:

  * Any regular or prescribed use of opioid analgesics in the past 3 months.
  * Use of prescription or OTC medications known to interact with alcohol within 2 weeks of the study. These include, but may not be limited to: isosorbide, nitroglycerine, benzodiazepines, warfarin, anti-depressants such as amitriptyline, clomipramine and nefazodone, anti-diabetes medications such as glyburide, metformin and tolbutamide, H2-antagonists for heartburn such as cimetidine and ranitidine, muscle relaxants, anti-epileptics including phenytoin and phenobarbital codeine, opioid analgesics including darvocet, percocet and hydrocodone, cough-and-cold preparations which contain anti-histamines, pain medicines and anti-inflammatories such as aspirin, ibuprofen, acetaminophen, celecoxib and naproxen.
  * Use of medications known to inhibit or induce enzymes that metabolize alcohol for 4 weeks prior to the study. These include chlorzoxazone, isoniazid, metronidazole and disulfiram.
  * Use of drugs known to affect hemodynamic response. These include antihypertensives, insulin and thyroid medications. [assessment: medical history and physical exam].
* Exclusion criteria for MRI:

  * Presence of ferromagnetic objects in the body that are contraindicated for MRI of the head (including but not limited to pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips, metallic prostheses, permanent eyeliner, implanted delivery pump, or shrapnel fragments).
  * Fear of enclosed spaces.
  * Inability to lie comfortable on back for up to 2 hours in the MRI scanner [assessment: NIAAA MRI Safety Screening Questionnaire].
* Exclusion criteria for women:

  * Pregnant [assessment: urine beta-hCG test at screening]. Women must also test negative on urine beta-hCG test at the start of every study visit.
  * Breast-feeding [assessment: medical history and physical exam].

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2016-06-08 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
Nalmefene-induced BOLD signal changes in neural regions associated with alcohol reward processing, including ventral striatum, amygdala, and insula | Post-administration
  functional MRI measure of brain activation.
Nalmefene-induced changes in IV alcohol self-administration | Post-administration
  human laboratory alcohol consumption measure.

SECONDARY OUTCOMES:
Nalmefene-induced BOLD signal changes in neural processing of aversive stimuli during fMRI | Post-adminstration
  functional MRI measure of brain activation.
Genotypic modulation (at the OPRM1 118 location) of Nalmafene's effects on primary outcome measures (BOLD signal change during alcohol reward processing and IV alcohol self-administration). | Post-administration
  human laboratory alcohol consumption measure.

CONTACTS AND LOCATIONS:
Overall Officials: Vijay A Ramchandani, Ph.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Gowin JL, Sloan ME, Kirk-Provencher KT, Rosenblatt SL, Penner AE, Stangl BL, Byrd ND, Swan JE, Ramchandani VA. Opioid receptor antagonism and neural response to monetary rewards: Pilot studies in light and heavy alcohol users. J Psychopharmacol. 2023 Sep;37(9):937-941. doi: 10.1177/02698811231191707. Epub 2023 Aug 2. PMID 37530456
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-AA-0037.html